CLINICAL TRIAL: NCT05411289
Title: The Effect of Acupressure on Labor Pain and Anxiety Levels During Labor in Primiparas Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona Mohamed Taha, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: P.T.REC/012/003704
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupressure (Experimental): Pressures were applied on three points consecutively, firstly on two points bilaterally Hugo point (LI4) and He-7 (Shenmen), then pressure was applied on sanyinjiao (SP6)
  Interventions: Procedure: acupressure
- sham acupressure (Sham Comparator)
  Interventions: Procedure: sham acupressure

INTERVENTIONS:
Procedure: acupressure — Pressures were applied on three points consecutively, firstly on two points bilaterally Hugo point (LI4) and He-7 (Shenmen), then pressure was applied on sanyinjiao (SP6).
  pressure was applied gradually for 30 seconds on the above mentioned points. Then this pressure was slowly intensified to the extent that the patient felt tingling, numbness, heaviness, and strain in the surrounding area.
  Arms: acupressure
Procedure: sham acupressure — Pressures were applied on sham points consecutively
  Arms: sham acupressure

SUMMARY:
the effect of acupressure on labor pain and anxiety levels during labor in primiparas women

ELIGIBILITY:
Inclusion Criteria:

* Primiparas women aged from 20 to 30 years old,
* gestational age of between 37 and 40 weeks according to ultrasonography.
* A fetal weight of between 2500 and 3500 g according to ultrasonography or clinical examination .
* They are transferred to labor room if active labor is in progress (defined as cervical dilatation 3 cm and the presence of regular uterine contraction,
* having a single and healthy fetus in the vertex position

Exclusion Criteria:

* who were needing an emergency C-section.
* Women having a current or previous high-risk pregnancy
* who have experienced pregnancy complications
* Women with a systemic disease during pregnancy . Women with a psychological disorder

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Anxiety level | about one hour
  To measure anxiety, the Spiberger inventory questionnaire will be used
labor pain | about one hour
  labor pain will be assessed using visual analogue scale.
  . It employs a 10-cm ruler scale with no pain sign at one end and the most intense pain sign at the other to allow users to assess their own pain

SECONDARY OUTCOMES:
pulse rate response | about one hour
  will measured using pulse oximetry
blood pressure response | about one hour
  will measured using sphygmomanometer

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hasanin ME, Elsayed SH, Taha MM. Effect of Acupressure on Anxiety and Pain Levels in Primiparous Women During Normal Labor: A Randomized Controlled Trial. J Integr Complement Med. 2024 Jul;30(7):654-661. doi: 10.1089/jicm.2023.0072. Epub 2023 Dec 20. PMID 38117578